CLINICAL TRIAL: NCT05655819
Title: A Randomized, Placebo-Controlled Trial Assessing the Effect of Glutamine on Intestinal Permeability and Symptoms in Patients With Functional Dyspepsia
Brief Title: A Study of Glutamine to Treat Intestinal Permeability in Functional Dyspepsia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David J. Cangemi (Other)
Responsible Party: Sponsor-Investigator, David J. Cangemi, Regulatory Sponsor and Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-004343
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glutamine Group (Active Comparator): Subjects will receive glutamine for 28 days.
  Interventions: Drug: Glutamine
- Placebo Group (Placebo Comparator): Subjects will receive placebo for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glutamine — 5 gram powder, one rounded teaspoon, dissolved in 8 ounces of water or juice prior to drinking) taken orally three times per day
  Arms: Glutamine Group
Drug: Placebo — Lactose powder dissolved in 8 ounces of water or juice prior to drinking, taken orally three times per day. Looks exactly like the study drug, but it contains no active ingredient.
  Arms: Placebo Group

SUMMARY:
The purpose of this research is to collect data from patients diagnosed with functional dyspepsia who are treated with glutamine and describe safety and treatment results compared to patients taking a placebo. Glutamine, an essential amino acid in humans, is an important energy source for cells lining the gastrointestinal tract and has been shown to play an important role in regulating the strength of the intestinal wall.

ELIGIBILITY:
Inclusion Criteria:

* Meet Rome IV criteria for functional dyspepsia (https://theromefoundation.org/rome-iv/rome-iv-criteria/)
* Patients will generally be in good health. During initial evaluation, patients' symptoms will be assessed and patients categorized into either the PDS, EPS or mixed subtype of FD.

Exclusion Criteria:

* Significant comorbid illness
* Symptoms are thought to represent an organic disorder (e.g., peptic ulcer disease, hepatitis, pancreatitis, inflammatory bowel disease, type I diabetes, a known malignancy, radiation-induced injury, an active infection, vasculitis, celiac disease), or if the patients have known esophagitis, eosinophilic esophagitis or H. pylori.
* Prior surgery to the esophagus, stomach or duodenum will be excluded, as will those taking proton pump inhibitors (PPIs), opioids, corticosteroids and those taking regular (daily) antihistamines, non-steroidal anti-inflammatory drugs (NSAIDs), or mast-cell stabilizing agents within the prior 2 weeks. Of note, patients taking PPIs will be given the opportunity to discontinue their PPI in favor of famotidine 20 mg daily for 2 weeks before enrollment.
* Known allergies to lactulose: mannitol.
* Active tobacco use and excessive alcohol use (defined as 8 or more drinks per week for women or 15 or more drinks per week for men; http://ww.cdc.gov)
* Co-existing IBS will be allowed to enter the study as long as symptoms are not predominant.
* Hepatic and renal impairment within the past 6 months. Defined as AST/ALT > 2X ULN, Total Bilirubin > 2 X ULN, Estimated Glomerular Filtration Rate (eGFR) of < 60 mL/min/BSA.
* Diagnosed with galactosemia.
* Pregnant or breastfeeding women.
* Patients with documented or reported lactose intolerance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Functional Dyspepsia symptoms | Baseline, 4 weeks
  Assessed by the validated self-reported Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) questionnaire total score. 20-item questionnaire measuring severity of symptoms related to gastrointestinal problem on scale from 0 = no symptoms to 5=very severe. Total score range 0-100 with higher score indicating greater severity of gastrointestinal symptoms.
Change in symptoms of bloating | Baseline, 4 weeks
  Assessed by the validated self-reported Mayo Bloating questionnaire (MBQ). 45-item questionnaire to describe symptoms of bloating and distension.
Changes in small bowel intestinal permeability | Baseline, 4 weeks
  Assessed using the validated lactulose: mannitol urine test
Adverse Events | 4 weeks
  Number of adverse events (serious and non-serious) reported

CONTACTS AND LOCATIONS:
Overall Officials: David Cangemi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Torsak Vimoktayon, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials